CLINICAL TRIAL: NCT06508320
Title: A Phase 2, Randomized, Observer-blind Study to Evaluate the Safety, Reactogenicity, and Immunogenicity in Relation to the Product Attributes of mRNA-1083 (SARS-CoV-2 and Influenza) Vaccine in Adults ≥50 to <65 Years of Age
Brief Title: A Clinical Study to Investigate the Safety and Immunogenicity in Relation to Product Attributes of mRNA-1083 (Severe Acute Respiratory Syndrome Coronavirus 2 [SARS-CoV-2] and Influenza Vaccine)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: mRNA-1083-P201
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Influenza; SARS-CoV-2
Keywords: Influenza; SARS-CoV-2; mRNA-1083
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 Group 1: mRNA-1083 Lot A (Experimental): Participants will receive mRNA-1083 Lot A as a single injection on Day 1 in Part 1.
  Interventions: Biological: mRNA-1083
- Part 1 Group 2: mRNA-1083 Lot B (Experimental): Participants will receive mRNA-1083 Lot B as a single injection on Day 1 in Part 1.
  Interventions: Biological: mRNA-1083
- Part 1 Group 3: mRNA-1083 Lot C (Experimental): Participants will receive mRNA-1083 Lot C as a single injection on Day 1 in Part 1.
  Interventions: Biological: mRNA-1083
- Part 1 Group 4: mRNA-1083 Lot D (Experimental): Participants will receive mRNA-1083 Lot D as a single injection on Day 1 in Part 1.
  Interventions: Biological: mRNA-1083
- Part 2 Group 5: mRNA-1083 Lot A (Experimental): Participants will receive mRNA-1083 Lot A as a single injection on Day 1 in Part 2.
  Interventions: Biological: mRNA-1083
- Part 2 Group 6: mRNA-1083 Lot E (Experimental): Participants will receive mRNA-1083 Lot E as a single injection on Day 1 in Part 2.
  Interventions: Biological: mRNA-1083

INTERVENTIONS:
Biological: mRNA-1083 — IM injection in a deltoid muscle.

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity, and immunogenicity in relation to the product attributes of mRNA-1083 vaccine when administered as a single intramuscular (IM) injection in adults ≥50 to <65 years of age.

DETAILED DESCRIPTION:
The study will be comprised of 2 parts, Parts 1 and 2. In Part 1, participants will be randomized into 4 study groups (Lots A, B, C, and D). Upon completion of Part 1, participants will be randomized into 2 study groups (Lots A and E) in Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Investigator assessment that the participant understands and is willing and physically able to comply with protocol-mandated follow-up, including all procedures.
2. Participants of nonchildbearing potential may be enrolled in the study.
3. Participants who could become pregnant: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy.
4. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
5. Have received an influenza vaccine in the previous season (since September 2023 for Part 1, since Sep 2024 for Part 2).

Exclusion Criteria:

1. Reported diagnosis or condition that is associated with increased risk of severe influenza disease or complications, including individuals with chronic medical conditions.
2. Reported history of congenital or acquired immunodeficiency, immunosuppressive condition, asplenia, or recurrent severe infections.
3. History of anaphylaxis or severe hypersensitivity reaction requiring medical intervention after receipt of any of the following: mRNA vaccine or therapeutic; components of an mRNA vaccine or therapeutic; influenza vaccine; or components of an influenza vaccine, including egg protein.
4. Received corticosteroids at ≥10 milligrams (mg)/day of prednisone or equivalent for >14 days in total within 90 days prior to Day 1 or is anticipating the need for corticosteroids at any time during the study.
5. Received systemic immunosuppressive treatment, including long-acting biological therapies that affect immune responses (e.g., infliximab), within 180 days prior to Day 1 or plans to do so during the study.
6. Received or plans to receive any vaccine authorized or approved by a local health agency within 28 days prior to Day 1 or plans to do so within 28 days post study injection.
7. Received a licensed seasonal influenza vaccine within 150 days prior to Day 1.
8. Received a licensed/authorized SARS-CoV-2 vaccine within 90 days prior to Day 1.
9. Received any investigational influenza vaccine, investigational coronavirus disease 2019 (COVID-19) vaccine, or investigational combination vaccine for influenza and COVID-19 within 12 months prior to Day 1. Participants from mRNA-1083-P201 Part 1 will also be excluded from Part 2.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 932 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Value of Antibodies at Day 29, as Measured by Hemagglutinin Inhibition (HAI) Assay for Influenza | Day 29
Geometric Mean Value of Antibodies at Day 29, as Measured by Pseudovirus Neutralization Assay (PsVNA) for SARS-CoV-2 | Day 29
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 7 (7 days after vaccination)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 28 (28 days after vaccination)
Number of Participants with Medically Attended Adverse Events (MAAEs) | Up to Day 181
Number of Participants with Adverse Events of Special Interest (AESIs) | Up to Day 181
Number of Participants with Serious Adverse Events (SAEs) | Up to Day 181
Number of Participants with AEs Leading to Discontinuation from Study Participation | Up to Day 181

SECONDARY OUTCOMES:
Geometric Mean Fold Rise (GMFR) of Antibodies at Day 29 Relative to Day 1, as Measured by HAI Assay for Influenza | Day 1, Day 29
GMFR of Antibodies at Day 29 Relative to Day 1, as Measured by PsVNA for SARS-CoV-2 | Day 1, Day 29
Seroconversion Rate (SCR) in Anti-hemagglutinin (HA) Antibody Values at Day 29, as Measured by HAI Assay for Influenza | Day 29
Seroresponse Rate (SRR) in Neutralizing Antibody (nAb) Values at Day 29, as Measured by PsVNA for SARS-CoV-2 | Day 29

CONTACTS AND LOCATIONS:
Locations (16):
- United States (12):
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Cenexel RCA, Hollywood, Florida
  - Suncoast Research Group, LLC DBA Flourish Research, Miami, Florida
  - Cenexel IRA, Decatur, Georgia
  - DM Clinical Research - River Forest, River Forest, Illinois
  - JCCT, Lenexa, Kansas
  - Hassman Research Institute - Berlin - CenExel - PPDS, Marlton, New Jersey
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - DM Clinical Research - Cyfair Clinical Research Center - PPDS, Houston, Texas
  - Clinical Trials of Texas, LLC DBA Flourish Research, San Antonio, Texas
  - DM Clinical Research - Sugarland, Sugar Land, Texas
  - DM Clinical Research - Tomball MDC, Tomball, Texas
- Canada (4):
  - Centricity Research, Toronto, Ontario
  - Centricity Research, Pointe-Claire, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - Diex Recherche Québec Inc., Québec